CLINICAL TRIAL: NCT03694275
Title: A Multicenter, Open-label, Pilot Study of TAK-935 (OV935) in Patients With 15Q Duplication Syndrome or CDKL5 Deficiency Disorder (ARCADE Study)
Brief Title: A Multicenter, Open-label, Pilot Study of Soticlestat (TAK-935/OV935) in Participants With 15Q Duplication Syndrome (Dup 15q) or Cyclin-Dependent Kinase-Like 5 (CDKL5) Deficiency Disorder (ARCADE STUDY)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Collaborators: Healx AI (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-935-18-002 (OV935); U1111-1219-5787 (Registry Identifier: WHO); 2022-001315-44 (EudraCT Number)
Record Dates: First submitted 2018-09-27; First posted 2018-10-03 (Actual); Results first posted 2021-04-20 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: 15q Duplication Syndrome; CDKL5 Deficiency Disease
Keywords: Drug Therapy; 15q Duplication Syndrome (Dup15q); CDKL5 Deficiency Disorder (CDD); Brain Diseases; Epilepsy; Central Nervous System Diseases; Autism; Cholesterol 24S-hydroxylase inhibitor; Anti-epilepsy drug; Anticonvulsants
MeSH Terms: conditions — Polyposis Syndrome, Hereditary Mixed, 1; CDKL5 deficiency disorder; Brain Diseases; Epilepsy; Central Nervous System Diseases; Autistic Disorder | interventions — soticlestat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Soticlestat Dup 15q (Experimental): Soticlestat tablets twice daily (BID) orally or via gastrostomy tube (G-tube)/ percutaneous endoscopic gastrostomy (PEG) tube, BID. Participants with Dup 15q weighing <60 kg at Baseline received total daily dose of study drug calculated based on body weight. Participants weighing ≥60 kg at Baseline, were administered with 200 mg/day followed by 400 mg/day, then 600 mg/day, up to Week 20.
  Interventions: Drug: Soticlestat
- Soticlestat CDD (Experimental): Soticlestat tablets BID orally or via G-tube/ PEG tube, BID. Participants with CDD weighing <60 kg at Baseline received total daily dose of study drug calculated based on body weight. Participants weighing ≥60 kg at Baseline, were administered with 200 mg/day followed by 400 mg/day, then 600 mg/day, up to Week 20.
  Interventions: Drug: Soticlestat

INTERVENTIONS:
Drug: Soticlestat — TAK-935 tablets
  Other Names: TAK-935

SUMMARY:
The purpose of this study is to investigate the effect of soticlestat on the frequency of motor seizures for participants with Dup15q or CDD during the Maintenance Period.

DETAILED DESCRIPTION:
The drug being tested in this study is called soticlestat. Soticlestat is being tested to treat people with Dup 15q or CDD. This study will assess the effects of TAK-935 on seizure frequency, safety.

The study will enroll approximately 30 participants. Participants will be enrolled into 2 groups based on their diagnosis as: Dup 15q or CDD.

All participants will be asked to take soticlestat tablets twice daily with or without food.

The study comprises of 2 periods: Screening/Baseline Period and Treatment Period (Dose Optimization and Maintenance). The overall time to participate in this study is approximately 30 weeks, including 4 to 6 weeks Screening/Baseline Period, 20 weeks Treatment Period, 2 weeks Taper, and 2 weeks safety follow up period. Participants completing this study will have an option to enroll in the open-label extension (OLE) study, under a separate protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of Dup 15q or CDKL5 deficiency disorder.
2. Currently taking 1 to 6 antiepileptic drugs (AEDs) at a stable dose.

Exclusion Criteria:

1. Two or more episodes of convulsive status epilepticus per 3 months requiring hospitalization and intubation.
2. Currently receiving a study drug or participated in a clinical study involving another investigational product in the previous month.

Ages: 2 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2020-07-13 (Actual); Study Completion 2020-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (8):
- United States (8):
  - UCLA, Los Angeles, California
  - Research Institute Children's Hospital Colorado, Aurora, Colorado
  - Center for Rare Neurological Diseases, Norcross, Georgia
  - Center for Rare Neurological Diseases (CRND)--Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital Translational Neuroscience Center, Boston, Massachusetts
  - Minnesota Epilepsy Group, P.A., Saint Paul, Minnesota
  - New York University (NYU), New York, New York
  - Columbia University Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Demarest S, Jeste S, Agarwal N, Arkilo D, Asgharnejad M, Hsiao S, Thibert R. Efficacy, safety, and tolerability of soticlestat as adjunctive therapy for the treatment of seizures in patients with Dup15q syndrome or CDKL5 deficiency disorder in an open-label signal-finding phase II study (ARCADE). Epilepsy Behav. 2023 May;142:109173. doi: 10.1016/j.yebeh.2023.109173. Epub 2023 Apr 1. PMID 37011526

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 8 investigative sites in the United States from 10 September 2018 to 31 July 2020.
Pre-assignment Details: Participants with a diagnosis of 15q duplication syndrome (Dup15q) or CDKL5 deficiency disorder (CDD) were enrolled in 2 cohorts to receive treatment with TAK-935 for up to 20 weeks Treatment Period (8-week Dose Optimization Period and 12-week Maintenance Period).
Groups:
- Soticlestat Dup15q: Soticlestat tablets twice daily (BID) orally or via gastrostomy tube (G-tube)/ percutaneous endoscopic gastrostomy (PEG) tube, BID. Participants with Dup15q weighing <60 kg at Baseline received total daily dose of study drug calculated based on body weight. Participants weighing ≥60 kg at Baseline, were administered with 200 mg/day followed by 400 mg/day, then 600 mg/day, up to Week 20.
Period: Overall Study
Arm/Group | Soticlestat Dup15q | Soticlestat CDD
Started | 8 | 12
Completed | 8 | 10
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Reason not Specified | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who have received at least 1 dose of study drug.
Groups:
- Soticlestat Dup15q: Soticlestat tablets BID orally or via G-tube/ PEG tube, BID. Participants with Dup15q weighing <60 kg at Baseline received total daily dose of study drug calculated based on body weight. Participants weighing ≥60 kg at Baseline, were administered with 200 mg/day followed by 400 mg/day, then 600 mg/day, up to Week 20.
- Total: Total of all reporting groups
Arm/Group | Soticlestat Dup15q | Soticlestat CDD | Total
Number analyzed (Participants) | 8 | 12 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.4 (6.00) | 7.6 (5.30) | 10.7 (6.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 9 | 12
  Male | 5 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 12 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 11 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 12 | 20
Height [Mean (Standard Deviation); unit: cm] | 148.54 (14.965) | 124.59 (26.882) | 134.17 (25.412)
Weight [Mean (Standard Deviation); unit: kg] | 43.40 (13.678) | 26.28 (12.511) | 33.13 (15.283)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI= weight (kg)/height (m^2).
  kg/m^2 | 19.21 (4.149) | 16.00 (1.874) | 17.28 (3.314)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Motor Seizure Frequency Per 28 Days During the Maintenance Period
Description: Seizure frequency per 28 days is defined as total number of Seizures reported during the period divided by number of days with no missing seizure count during the period multiplied by 28. Percent Change from Baseline is defined as (frequency of seizures per 28 days during maintenance period - frequency of seizures per 28 days at Baseline) divided by frequency of seizures per 28 days at Baseline multiplied by 100. Positive percent change from Baseline indicates seizure increase and negative percent change from Baseline indicates seizure decrease.
Time Frame: Maintenance Period: Weeks 9 to 20
Population: Modified Intent-to-Treat (mITT) Analysis Set included all participants who have received at least 1 dose of study drug and have been assessed for at least 1 day in the Treatment Period. Overall number analyzed are the number of participants with data available for analyses.
Measure: Median (Full Range); unit: percent change
Arm/Group | Soticlestat Dup15q | Soticlestat CDD
Number analyzed (Participants) | 8 | 11
percent change | 11.7 [-90 to 39] | -23.6 [-100 to 107]

2. Secondary Outcome: Percent Change From Baseline in Motor Seizure Frequency Per 28 Days During the Treatment Period
Description: Seizure frequency per 28 days is defined as total number of Seizures reported during the period divided by number of days with no missing seizure count during the period multiplied by 28. Percent Change from Baseline is defined as (frequency of seizures per 28 days during the treatment period - frequency of seizures per 28 days at Baseline) divided by frequency of seizures per 28 days at Baseline multiplied by 100. Positive percent change from Baseline indicates seizure increase and negative percent change from Baseline indicates seizure decrease.
Time Frame: Treatment Period: Weeks 0 to 20
Population: mITT Analysis Set included all participants who have received at least 1 dose of study drug and have been assessed for at least 1 day in the Treatment Period.
Measure: Median (Full Range); unit: percent change
Arm/Group | Soticlestat Dup15q | Soticlestat CDD
Number analyzed (Participants) | 8 | 12
percent change | 13.4 [-89 to 30] | -13.6 [-93 to 48]

3. Secondary Outcome: Percentage of Participants Considered as Treatment Responders During the Maintenance Period
Description: Responders are defined as having over 50% motor seizure reduction compared to Baseline. Percent reduction from Baseline (%) is defined as [(Maintenance Period motor Seizure Frequency - Baseline Period motor Seizure Frequency) divided by Baseline motor Seizure Frequency] multiplied by 100. Data is reported as reduction of 25%, 50%, 75% and 100% or more in motor seizures from Baseline.
Time Frame: Maintenance Period: Weeks 9 to 20
Population: mITT Analysis Set included all participants who have received at least 1 dose of study drug and have been assessed for at least 1 day in the Treatment Period. Overall number analyzed is the number of participants with data available for analyses.
Measure: Number; unit: percentage of participants
Arm/Group | Soticlestat Dup15q | Soticlestat CDD
Number analyzed (Participants) | 8 | 11
percentage of participants
  <=0% Reduction | 62.5 | 27.3
  >0% to <25% Reduction | 12.5 | 27.3
  >=25% to <50% Reduction | 12.5 | 18.2
  >=50% to <75% Reduction | 0 | 18.2
  >=75% to 100% Reduction | 12.5 | 9.1

4. Secondary Outcome: Percent Change From Baseline in Frequency of Motor Seizures Longer Than 5 Minutes in Participants With CDD
Description: Seizure frequency is defined as total number of Seizures reported during the period divided by number of days with no missing seizure count during the period. Percent Change from Baseline is defined as (frequency of seizures during Treatment period - frequency of seizures at Baseline) divided by frequency of seizures at Baseline multiplied by 100. Positive percent change from Baseline indicates seizure increase and negative percent change from Baseline indicates seizure decrease. The data is reported only for CDD participants.
Time Frame: Treatment Period: Weeks 0 to 20
Population: mITT Analysis Set included all participants who have received at least 1 dose of study drug and have been assessed for at least 1 day in the Treatment Period. Overall number analyzed are all participants whose analyses were conducted using observed values and no imputation was done for missing data.
Measure: Median (Full Range); unit: percent change
Arm/Group | Soticlestat CDD
Number analyzed (Participants) | 6
percent change | -54.0 [-86 to 11]

5. Secondary Outcome: Proportion of Motor Seizure-free Days in Participants During the Maintenance Period
Description: Seizure-free days is defined as number of days with zero motor seizure during the period the Maintenance Period divided by number of days participant was in the Maintenance Period.
Time Frame: Maintenance Period: Weeks 9 to 20
Population: as for outcome 3
Measure: Median (Full Range); unit: days/28 days
Arm/Group | Soticlestat Dup15q | Soticlestat CDD
Number analyzed (Participants) | 8 | 11
days/28 days | 0.1 [0 to 1] | 0.1 [0 to 1]

6. Secondary Outcome: Change From Baseline in Clinician's Global Impression of Severity (CGI-S) Responses of Investigator
Description: The CGI-S focuses on clinician's observations of the participant's cognitive, functional, and behavioral performance since the beginning of the study. The CGI-S is rated on a 7-point scale, with the severity of illness scale using a range of responses where, 1= normal, not at all ill, 2= borderline mentally ill, 3= mildly ill, 4= moderately ill, 5= markedly ill, 6= severely ill and 7=amongst the most extremely ill participants. Negative change from Baseline indicates improvement.
Time Frame: Baseline to Week 20
Population: mITT Analysis Set included all participants who have received at least 1 dose of study drug and have been assessed for at least 1 day in the Treatment Period. Number analyzed is the number of participants with data available for analyses at the given timepoint.
Measure: Median (Full Range); unit: score on scale
Arm/Group | Soticlestat Dup15q | Soticlestat CDD
Number analyzed (Participants) | 8 | 12
score on scale
  Baseline | 5.0 [4 to 6] | 5.0 [4 to 6]
  Change From Baseline at Week 20: number analyzed (Participants) | 6 | 12
  Change From Baseline at Week 20 | 0.0 [-2 to 0] | 0.0 [-1 to 1]

7. Secondary Outcome: Percentage of Participants With Clinical Global Impression of Change (CGI-C) Responses as Per the Investigator Reported Impression
Description: CGI-Change (CGI-C) treatment response ratings should take account of both therapeutic efficacy and treatment-related AEs. Each component of the CGI is rated separately; the instrument does not yield a global score. The CGI-C is rated on a 5-point scale, where, 0 = marked improvement and no side-effects, 1 = marked improvement and minimal side-effects, 2 = no change, 3 = minimal improvement and marked side-effects and 4 = unchanged or worse and side-effects outweigh the therapeutic effect. Lower scores indicated improvement.
Time Frame: Week 20
Population: mITT Analysis Set included all participants who have received at least 1 dose of study drug and have been assessed for at least 1 day in the Treatment Period. Overall number analyzed is the number of participants with data available for analyses at given timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Soticlestat Dup15q | Soticlestat CDD
Number analyzed (Participants) | 6 | 12
percentage of participants
  Week 20, Score 0 | 33.3 | 33.3
  Week 20, Score 1 | 0 | 33.3
  Week 20, Score 2 | 50.0 | 33.3
  Week 20, Score 3 | 16.7 | 0
  Week 20, Score 4 | 0 | 0

8. Secondary Outcome: Percentage of Participants With Care Clinical Global Impression of Change (CGI-C) Responses of Parent/Family
Description: CGI-Change (CGI-C) treatment response ratings should take account of both therapeutic efficacy and treatment-related AEs. Each component of the CGI is rated separately; the instrument does not yield a global score. The CGI-C is rated on a 7-point scale where, 1 = very much improved, 2 = much improved, 3 = slightly improved, 4= no change, 5= slightly worse, 6= much worse and 7= very much worse and marked side-effects. Lower scores indicated improvement.
Time Frame: Week 20
Population: mITT Analysis Set included all participants who have received at least 1 dose of study drug and have been assessed for at least 1 day in the Treatment Period. Overall number analyzed is the number of participants with data available for analyses at the given timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Soticlestat Dup15q | Soticlestat CDD
Number analyzed (Participants) | 6 | 12
percentage of participants
  Week 20, Score 1 | 0 | 16.7
  Week 20, Score 2 | 16.7 | 25.0
  Week 20, Score 3 | 33.3 | 50.0
  Week 20, Score 4 | 50.0 | 0
  Week 20, Score 5 | 0 | 8.3
  Week 20, Score 6 | 0 | 0
  Week 20, Score 7 | 0 | 0

9. Secondary Outcome: Change From Baseline of Plasma 24S-hydroxycholesterol (24HC) Levels
Time Frame: Baseline to Week 20
Population: mITT Analysis Set included all participants who have received at least 1 dose of study drug and have been assessed for at least 1 day in the Treatment Period. Overall number analyzed is the number of participants with data available for analyses. Number analyzed is the number of participants with data available for analyses at the given timepoint.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Soticlestat Dup15q | Soticlestat CDD
Number analyzed (Participants) | 8 | 11
ng/mL
  Baseline | 57.08 (24.195) | 115.29 (73.587)
  Change from Baseline at Week 20: number analyzed (Participants) | 4 | 5
  Change from Baseline at Week 20 | -34.71 (16.578) | -75.64 (29.284)

10. Secondary Outcome: Change From Baseline in Seizure Frequency in Participants Treated With TAK-935 as an Adjunctive Therapy
Description: Seizure Frequency per 28 days is defined as total number of Seizures reported during the period divided by number of days with no missing seizure during the period seizures were assessed multiplied by 28. Positive change from Baseline indicates seizure increase and negative change from Baseline indicates seizure decrease.
Time Frame: Baseline to Week 20
Population: as for outcome 2
Measure: Median (Full Range); unit: seizures per 28 days
Arm/Group | Soticlestat Dup15q | Soticlestat CDD
Number analyzed (Participants) | 8 | 12
seizures per 28 days
  Baseline | 128.4 [35 to 224] | 77.8 [10 to 374]
  Change From Baseline | 13.2 [-31 to 67] | -3.4 [-210 to 28]

ADVERSE EVENTS:
Time Frame: From the first dose to 30 days post-last dose of study treatment (Up to 24 weeks)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Soticlestat Dup15q | Soticlestat CDD
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/8 | 2/12
Other Adverse Events (participants affected / at risk) | 7/8 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Soticlestat Dup15q (N=8) | Soticlestat CDD (N=12)
Anaphylactic reaction (Immune system disorders) | 1 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Soticlestat Dup15q (N=8) | Soticlestat CDD (N=12)
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 4
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 2 | 0
Asthenia (General disorders) | 0 | 1
Peripheral swelling (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 1
Ear infection (Infections and infestations) | 0 | 2
Nasopharyngitis (Infections and infestations) | 1 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Face injury (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Blood bicarbonate decreased (Investigations) | 0 | 2
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0
Anticonvulsant drug level increased (Investigations) | 1 | 0
Blood cholesterol increased (Investigations) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1
Blood triglycerides increased (Investigations) | 0 | 1
C-reactive protein increased (Investigations) | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 1
Electrocardiogram ST-T change (Investigations) | 0 | 1
Haematocrit increased (Investigations) | 0 | 1
International normalised ratio increased (Investigations) | 1 | 0
Low density lipoprotein increased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Oxygen saturation decreased (Investigations) | 0 | 1
Platelet count increased (Investigations) | 0 | 1
White blood cell count increased (Investigations) | 0 | 1
Seizure (Nervous system disorders) | 2 | 1
Lethargy (Nervous system disorders) | 2 | 0
Partial seizures (Nervous system disorders) | 0 | 2
Tonic convulsion (Nervous system disorders) | 0 | 2
Atonic seizures (Nervous system disorders) | 0 | 1
Balance disorder (Nervous system disorders) | 1 | 0
Drooling (Nervous system disorders) | 1 | 0
Hypersomnia (Nervous system disorders) | 1 | 0
Hypotonia (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Agitation (Psychiatric disorders) | 1 | 1
Initial insomnia (Psychiatric disorders) | 0 | 1
Irritability (Psychiatric disorders) | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 1
Neurogenic bladder (Renal and urinary disorders) | 0 | 1
Urinary retentio (Renal and urinary disorders) | 0 | 1
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2019-11-21): https://cdn.clinicaltrials.gov/large-docs/75/NCT03694275/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-25): https://cdn.clinicaltrials.gov/large-docs/75/NCT03694275/SAP_001.pdf